CLINICAL TRIAL: NCT00742547
Title: DIANA - Diabetes Mellitus: Neue Wege Der Optimierung Der allgemeinärztlichen Betreuung
Brief Title: Type 2 Diabetes Mellitus: New Approaches to Optimize Medical Care in General Practice
Acronym: DIANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Collaborators: Heidelberg University (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-r86/zoo8
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: prevention; health services research
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No telephone counseling + usual care
- Telephone Counseling (Experimental): Telephone counseling + usual care
  Interventions: Other: Telephone counseling

INTERVENTIONS:
Other: Telephone counseling — Telephone counseling is provided once a month by the medical secretary of the general practitioner's practices
  Arms: Telephone Counseling

SUMMARY:
Patients with type-2 diabetes mellitus have an higher risk developing secondary disorders. In an epidemiological longitudinal study of about 1.150 patients with type 2 diabetes mellitus we investigate determinants and predictors for long-term prognosis. The patients are recruited and supervised in practices of general practitioners of the administrative district of Ludwigsburg/Heilbronn (Baden-Württemberg, Germany). In a subgroup of about 200 patients with a dissatisfactory metabolic status (HbA1c > 7,5%) a randomised interventional study is performed. The intervention comprises a telephone counseling by the medical secretary of each practice executed in a predefined period of time. The outcome parameters of interest are the change of HbA1c, the development of secondary disorders and adverse events, quality of life and risk factor control, as well as hospitalization and mortality.

The aim of the study was to develop an patient-centred instrument implementable in the routine medical care in order to enhance the prognosis of patients with type-2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patient with type-2 diabetes mellitus attending the general practitioner's in the time from October to December 2008
* Ability to take part in the study

Exclusion Criteria:

* Nursing home resident
* Insufficient knowledge of the German language
* Palliative health care with limited life expectancy
* Emergency outpatient
* All outpatients who attend the general practitioner by way of exception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 18 months

SECONDARY OUTCOMES:
hospitalization | 18 month
CHD, mortality | 18 months
lipid metabolism control | 18 months
risk factor control (eg. body weight, physical activity, smoking) | 18 months
health-related quality of life | 18 months
incidence of diabetes-related complications | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Brenner, MD, MPH, Principal Investigator — German Cancer Research Center
Locations (37):
- Germany (37):
  - Christoph Lücke, MD, Beilstein, Baden-Wurttemberg
  - Andrea Walliser-Klöpfer, MD, Benningen am Neckar, Baden-Wurttemberg
  - Nader Heydari, MD, Fellbach, Baden-Wurttemberg
  - Adelheid Halttunen, MD, Gemmingen, Baden-Wurttemberg
  - Hans-Joachim Essich, MD, Heilbronn, Baden-Wurttemberg
  - Jürgen Wollweber, MD, Heilbronn, Baden-Wurttemberg
  - Volker Naser, MD, Heilbronn, Baden-Wurttemberg
  - Andreas Wößner, MD, Heilbronn, Baden-Wurttemberg
  - Ullrich Barthelmes, MD, Heilbronn, Baden-Wurttemberg
  - Axel Möller, MD, Heilbronn, Baden-Wurttemberg
  - Miroslaw Wyszynski, MD, Heilbronn, Baden-Wurttemberg
  - Ulrich Hofmann, MD, Ilsfeld-Auenstein, Baden-Wurttemberg
  - Hans Martin Schweizer, MD, Korntal, Baden-Wurttemberg
  - Eberhard Rieker, MD, Lauffen am Neckar, Baden-Wurttemberg
  - Bernd Leuchs, MD, Leonberg, Baden-Wurttemberg
  - Gerhard Günther, MD, Leonberg, Baden-Wurttemberg
  - Thomas Baartz, MD, Leonberg, Baden-Wurttemberg
  - Monika Muhler, MD, Löwenstein, Baden-Wurttemberg
  - Ulrich Wagner, MD, Ludwigsburg, Baden-Wurttemberg
  - Martin Heinrich, MD, Ludwigsburg, Baden-Wurttemberg
  - Franz Lang, MD, Marbach am Neckar, Baden-Wurttemberg
  - Jürgen Wirth, MD, Marbach am Neckar, Baden-Wurttemberg
  - Alfred Preisner, MD, Massenbachhausen, Baden-Wurttemberg
  - Michael Spiel, MD, Murr, Baden-Wurttemberg
  - Hans-Jürgen Sommerer, MD, Neckarsulm, Baden-Wurttemberg
  - Dietmar Kunz, MD, Neckarsulm, Baden-Wurttemberg
  - Hartmut Jungjohann, MD, Neckarsulm, Baden-Wurttemberg
  - Jürgen Herbers, MD, Pleidelsheim, Baden-Wurttemberg
  - Ulf-Michael Werner, MD, Remshalden, Baden-Wurttemberg
  - Frank Röder, MD, Schwaikheim, Baden-Wurttemberg
  - Gisela Gramlich, MD, Untergruppenbach, Baden-Wurttemberg
  - Ildiko Tasic, Vaihingen-Enz, Baden-Wurttemberg
  - Karl Schütz, MD, Weinsberg, Baden-Wurttemberg
  - Sigmund Jakob, Weinsberg, Baden-Wurttemberg
  - Kurt Weber, MD, Weissach, Baden-Wurttemberg
  - Dietmar Zinßer, MD, Winnenden, Baden-Wurttemberg
  - Odilo Schnabel, MD, Zaberfeld, Baden-Wurttemberg

REFERENCES:
- [Derived] Mons U, Raum E, Kramer HU, Ruter G, Rothenbacher D, Rosemann T, Szecsenyi J, Brenner H. Effectiveness of a supportive telephone counseling intervention in type 2 diabetes patients: randomized controlled study. PLoS One. 2013 Oct 30;8(10):e77954. doi: 10.1371/journal.pone.0077954. eCollection 2013. PMID 24205043
- [Derived] Kramer HU, Raum E, Ruter G, Schottker B, Rothenbacher D, Rosemann T, Szecsenyi J, Brenner H. Gender disparities in diabetes and coronary heart disease medication among patients with type 2 diabetes: results from the DIANA study. Cardiovasc Diabetol. 2012 Jul 27;11:88. doi: 10.1186/1475-2840-11-88. PMID 22838970